CLINICAL TRIAL: NCT03396146
Title: Assay for the Pancreatic Polypeptide: an Help for Clinical Practice Guidelines in Classification of the Diabetes
Acronym: DIAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Cochin Hospital's Hormonology Laboratory (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: K160403J; 2017-A00612-51 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2017-11-17; First posted 2018-01-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Type1diabetes
Keywords: Pancreatic polypeptide; Type 1 diabetes; Chronic pancreatitis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Type1diabetes with exocrine pancreatic function insufficiency (Experimental): 12 ml total blood tubes volume Fecal sample
  Interventions: Other: 12 ml total blood tubes volume; Other: Fecal sample
- Type1diabetes without exocrine pancreatic function insuficienc (Experimental): 12 ml total blood tubes volume Fecal sample
  Interventions: Other: 12 ml total blood tubes volume; Other: Fecal sample
- Type 3c diabetes (Active Comparator): 12 ml total blood tubes volume Fecal sample
  Interventions: Other: 12 ml total blood tubes volume; Other: Fecal sample

INTERVENTIONS:
Other: 12 ml total blood tubes volume — 12 ml total blood tubes at 0, +60, + 90, + 120 minutes before and after a mixed meal
Other: Fecal sample — Fecal sample at inclusion

SUMMARY:
The purpose of this study is to evaluate global endocrine function within type 1 and type 3c diabetic patients, helping pancreatic polypeptide measurement.

DETAILED DESCRIPTION:
All diabetes are the result of endrocrine deficiency. The endocrine deficiency may be absolute, as in type 1 diabetes, considered as an elective and exclusive attack of pancreatic Beta cell, or it could be relative, as un type 2 diabetes.

More rarely, diabetes fit into a broader context of pancreatic failure, with diffuse involvement of the exocrine and endocrine function, suggesting an impairment of the whole endocrine secretion of the pancreas, affecting the entire islet of Langerhans, such as in type 3c diabetes, whose prototypes are total pancreatectomy, chronic alcoholic pancreatitis, cystic fibrosis.

The diagnostic of type 3c diabetes is not always obvious, with several clinical presentations, without biological specific disease tag. Moreover, it also appears that the common form of diabetes, type 1 and type 2, may be associated with an exocrine function deficit and with a decrease of the pancreatic volume correlated with exocrine function abnormalities, and a decrease of insulin secretion capacity. The consequences of a spread of the disease beyond the Beta cells remain uncertain, but they could be linked, as in type 3c diabetes, with severe form of hypoglycaemia, due to glucagon deficiency, or nutritional deficiency due to the exocrine deficiency.

The pancreatic polypeptide belongs to the neuropeptide Y family, it is produced by the endocrine pancreatic F cells, located in the hook and the head of the pancreas. Food intake stimulates its secretion. The role of the pancreatic polypeptide in human is uncertain.

Investigators propose to study the pancreatic polypeptide in type 1 and type 3c diabetes before and after a mixed meal in order to study the other endocrine functions of the islet of Langerhans, to evaluate the possibility, or not, of a more diffuse pancreatic involvement in type 1 diabetes, considered as an elective pathology of the pancreatic Beta cell.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients with type 1 diabetes with anti-GAD and / or IA2 and / or Znt8 positive antibodies, or characteristic clinical history, with and without exocrine deficiency (*)
* Patients with chronic alcoholic pancreatitis or cystic fibrosis origin (type 3c diabetes), complicated with diabetes defined by HbA1c> 6.5% or treated with oral anti-diabetic and / or insulin
* Patients who have given informed and written consent to participate in research
* Patients affiliated to a social security scheme (*): The exocrine deficiency is defined by an assay of fecal elastase:
* without deficit of exocrine function = fecal elastase = /> 100 μg / g
* with deficit of exocrine function = fecal elastase <100 μg / g

Exclusion Criteria:

* Pregnancy
* Severe renal impairment (eDFG <45 mL / min / 1.73 m²)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Measurement of pancreatic polypeptide for calculating the area under the curve | 1 day
  physiological parameters

SECONDARY OUTCOMES:
Measurement of C-peptide levels | 1 day
  physiological parameters
Measurement of fecal elastase level | at inclusion
  physiological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Etienne LARGER, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larger E, Philippe MF, Barbot-Trystram L, Radu A, Rotariu M, Nobecourt E, Boitard C. Pancreatic exocrine function in patients with diabetes. Diabet Med. 2012 Aug;29(8):1047-54. doi: 10.1111/j.1464-5491.2012.03597.x. PMID 22273174
- [Background] Philippe MF, Benabadji S, Barbot-Trystram L, Vadrot D, Boitard C, Larger E. Pancreatic volume and endocrine and exocrine functions in patients with diabetes. Pancreas. 2011 Apr;40(3):359-63. doi: 10.1097/MPA.0b013e3182072032. PMID 21283038
- [Background] Rickels MR, Bellin M, Toledo FG, Robertson RP, Andersen DK, Chari ST, Brand R, Frulloni L, Anderson MA, Whitcomb DC; PancreasFest Recommendation Conference Participants. Detection, evaluation and treatment of diabetes mellitus in chronic pancreatitis: recommendations from PancreasFest 2012. Pancreatology. 2013 Jul-Aug;13(4):336-42. doi: 10.1016/j.pan.2013.05.002. Epub 2013 May 17. PMID 23890130
- [Background] Khandekar N, Berning BA, Sainsbury A, Lin S. The role of pancreatic polypeptide in the regulation of energy homeostasis. Mol Cell Endocrinol. 2015 Dec 15;418 Pt 1:33-41. doi: 10.1016/j.mce.2015.06.028. Epub 2015 Jun 27. PMID 26123585
- [Background] Hennig R, Kekis PB, Friess H, Adrian TE, Buchler MW. Pancreatic polypeptide in pancreatitis. Peptides. 2002 Feb;23(2):331-8. doi: 10.1016/s0196-9781(01)00605-2. PMID 11825647
- [Background] Wang X, Zielinski MC, Misawa R, Wen P, Wang TY, Wang CZ, Witkowski P, Hara M. Quantitative analysis of pancreatic polypeptide cell distribution in the human pancreas. PLoS One. 2013;8(1):e55501. doi: 10.1371/journal.pone.0055501. Epub 2013 Jan 31. PMID 23383206
- [Background] Simonian HP, Kresge KM, Boden GH, Parkman HP. Differential effects of sham feeding and meal ingestion on ghrelin and pancreatic polypeptide levels: evidence for vagal efferent stimulation mediating ghrelin release. Neurogastroenterol Motil. 2005 Jun;17(3):348-54. doi: 10.1111/j.1365-2982.2004.00634.x. PMID 15916622
- [Background] Veedfald S, Plamboeck A, Hartmann B, Svendsen LB, Vilsboll T, Knop FK, Holst JJ. Pancreatic polypeptide responses to isoglycemic oral and intravenous glucose in humans with and without intact vagal innervation. Peptides. 2015 Sep;71:229-31. doi: 10.1016/j.peptides.2015.07.020. Epub 2015 Jul 26. PMID 26218807
- [Background] Batterham RL, Le Roux CW, Cohen MA, Park AJ, Ellis SM, Patterson M, Frost GS, Ghatei MA, Bloom SR. Pancreatic polypeptide reduces appetite and food intake in humans. J Clin Endocrinol Metab. 2003 Aug;88(8):3989-92. doi: 10.1210/jc.2003-030630. PMID 12915697
- [Background] Brunicardi FC, Chaiken RL, Ryan AS, Seymour NE, Hoffmann JA, Lebovitz HE, Chance RE, Gingerich RL, Andersen DK, Elahi D. Pancreatic polypeptide administration improves abnormal glucose metabolism in patients with chronic pancreatitis. J Clin Endocrinol Metab. 1996 Oct;81(10):3566-72. doi: 10.1210/jcem.81.10.8855802.
- [Background] Rabiee A, Galiatsatos P, Salas-Carrillo R, Thompson MJ, Andersen DK, Elahi D. Pancreatic polypeptide administration enhances insulin sensitivity and reduces the insulin requirement of patients on insulin pump therapy. J Diabetes Sci Technol. 2011 Nov 1;5(6):1521-8. doi: 10.1177/193229681100500629. PMID 22226275
- [Background] Henquin JC, Rahier J. Pancreatic alpha cell mass in European subjects with type 2 diabetes. Diabetologia. 2011 Jul;54(7):1720-5. doi: 10.1007/s00125-011-2118-4. Epub 2011 Apr 5. PMID 21465328
- [Background] Diedisheim M, Mallone R, Boitard C, Larger E. beta-cell Mass in Nondiabetic Autoantibody-Positive Subjects: An Analysis Based on the Network for Pancreatic Organ Donors Database. J Clin Endocrinol Metab. 2016 Apr;101(4):1390-7. doi: 10.1210/jc.2015-3756. Epub 2016 Feb 1. PMID 26829442
- [Background] Gerich JE, Langlois M, Noacco C, Karam JH, Forsham PH. Lack of glucagon response to hypoglycemia in diabetes: evidence for an intrinsic pancreatic alpha cell defect. Science. 1973 Oct 12;182(4108):171-3. doi: 10.1126/science.182.4108.171. PMID 4581053
- [Background] Lund A, Bagger JI, Wewer Albrechtsen NJ, Christensen M, Grondahl M, Hartmann B, Mathiesen ER, Hansen CP, Storkholm JH, van Hall G, Rehfeld JF, Hornburg D, Meissner F, Mann M, Larsen S, Holst JJ, Vilsboll T, Knop FK. Evidence of Extrapancreatic Glucagon Secretion in Man. Diabetes. 2016 Mar;65(3):585-97. doi: 10.2337/db15-1541. Epub 2015 Dec 15. PMID 26672094
- [Background] Tiengo A, Bessioud M, Valverde I, Tabbi-Anneni A, Delprato S, Alexandre J, Assan R. Absence of islet alpha cell function in pancreatectomized patients. Diabetologia. 1982 Jan;22(1):25-32. doi: 10.1007/BF00253865. PMID 6120875
- [Background] Haldorsen IS, Raeder H, Vesterhus M, Molven A, Njolstad PR. The role of pancreatic imaging in monogenic diabetes mellitus. Nat Rev Endocrinol. 2011 Nov 29;8(3):148-59. doi: 10.1038/nrendo.2011.197. PMID 22124438
- [Background] Bellanne-Chantelot C, Chauveau D, Gautier JF, Dubois-Laforgue D, Clauin S, Beaufils S, Wilhelm JM, Boitard C, Noel LH, Velho G, Timsit J. Clinical spectrum associated with hepatocyte nuclear factor-1beta mutations. Ann Intern Med. 2004 Apr 6;140(7):510-7. doi: 10.7326/0003-4819-140-7-200404060-00009. PMID 15068978
- [Background] Andersen BN, Hagen C, Klein HC, Stadil F, Worning H. Correlation between exocrine pancreatic secretion and serum concentration of human pancreatic polypeptide in chronic pancreatitis. Scand J Gastroenterol. 1980;15(6):699-704. doi: 10.3109/00365528009181517. PMID 7209380
- [Background] Matsumoto M, Wakasugi H, Ibayashi H. Plasma human pancreatic polypeptide response in chronic pancreatitis. Gastroenterol Jpn. 1982;17(1):25-30. doi: 10.1007/BF02774757. PMID 7042449
- [Background] Vu MK, Vecht J, Eddes EH, Biemond I, Lamers CB, Masclee AA. Antroduodenal motility in chronic pancreatitis: are abnormalities related to exocrine insufficiency? Am J Physiol Gastrointest Liver Physiol. 2000 Mar;278(3):G458-66. doi: 10.1152/ajpgi.2000.278.3.G458. PMID 10712266
- [Background] Sobngwi E, Boudou P, Mauvais-Jarvis F, Leblanc H, Velho G, Vexiau P, Porcher R, Hadjadj S, Pratley R, Tataranni PA, Calvo F, Gautier JF. Effect of a diabetic environment in utero on predisposition to type 2 diabetes. Lancet. 2003 May 31;361(9372):1861-5. doi: 10.1016/S0140-6736(03)13505-2. PMID 12788573
- [Background] Chia CW, Odetunde JO, Kim W, Carlson OD, Ferrucci L, Egan JM. GIP contributes to islet trihormonal abnormalities in type 2 diabetes. J Clin Endocrinol Metab. 2014 Jul;99(7):2477-85. doi: 10.1210/jc.2013-3994. Epub 2014 Apr 8. PMID 24712564
- [Background] Belinova L, Kahleova H, Malinska H, Topolcan O, Vrzalova J, Oliyarnyk O, Kazdova L, Hill M, Pelikanova T. Differential acute postprandial effects of processed meat and isocaloric vegan meals on the gastrointestinal hormone response in subjects suffering from type 2 diabetes and healthy controls: a randomized crossover study. PLoS One. 2014 Sep 15;9(9):e107561. doi: 10.1371/journal.pone.0107561. eCollection 2014. PMID 25222490
- [Background] Hart PA, Baichoo E, Bi Y, Hinton A, Kudva YC, Chari ST. Pancreatic polypeptide response to a mixed meal is blunted in pancreatic head cancer associated with diabetes mellitus. Pancreatology. 2015 Mar-Apr;15(2):162-6. doi: 10.1016/j.pan.2015.02.006. Epub 2015 Feb 24. PMID 25766398
- [Background] Sumithran P, Prendergast LA, Delbridge E, Purcell K, Shulkes A, Kriketos A, Proietto J. Long-term persistence of hormonal adaptations to weight loss. N Engl J Med. 2011 Oct 27;365(17):1597-604. doi: 10.1056/NEJMoa1105816. PMID 22029981
- [Background] Nealon WH, Townsend CM Jr, Thompson JC. The time course of beta cell dysfunction in chronic ethanol-induced pancreatitis: a prospective analysis. Surgery. 1988 Dec;104(6):1074-9. PMID 3057670
- [Background] Brunicardi FC, Druck P, Sun YS, Elahi D, Gingerich RL, Andersen DK. Regulation of pancreatic polypeptide secretion in the isolated perfused human pancreas. Am J Surg. 1988 Jan;155(1):63-9. doi: 10.1016/s0002-9610(88)80259-9. PMID 3277467
- [Result] Dehghani L, Bonnet-Serrano F, Abdul H, Alexandre-Heymann L, Guibourdenche J, Larger E. Pancreatic polypeptide in patients with type 1 diabetes and exocrine failure or chronic pancreatitis. The DIAPP study. Diabetes Metab. 2026 Jan;52(1):101712. doi: 10.1016/j.diabet.2025.101712. Epub 2025 Nov 9. PMID 41218735